CLINICAL TRIAL: NCT06947395
Title: VERIFI: A Multicenter, Case-Control Clinical Validation Study of the Multiplex Blood Protein Biomarker Test, PancreaSure, for Early Detection of Pancreatic Ductal Adenocarcinoma (PDAC) in High-Risk Patients
Brief Title: Clinical Validation of a Blood Biomarker Test to Detect Early-Stage Pancreatic Cancer (VERIFI)
Acronym: VERIFI
Status: Completed | Type: Observational
Sponsor: Immunovia, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: VERIFI-11
Record Dates: First submitted 2025-04-11; First posted 2025-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Cancer of the Pancreas; Pancreatic Cancer; Pancreas Neoplasms; Pancreatic Carcinoma Stage I; Pancreatic Carcinoma Stage II
Keywords: Early Detection of Cancer; Cancer Diagnostic; Early Detection of Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pancreatic Ductal Adenocarcinoma (PDAC) Stage I and Stage II Cases: PDAC case samples will be obtained from patients with newly diagnosed, treatment- naive PDAC (Stages I and II). PDAC cases will include patients with familial/genetic or sporadic disease identified by the institution or referred to it for clinical management.
  Interventions: Diagnostic Test: PancreaSure
- High-Risk Controls: Controls will consist of individuals who are at increased risk for PDAC because of their family history, known germline variants predisposing to PDAC, or the presence of pancreatic cystic lesions consistent with IPMNs. Note that cystic lesions between 1 and 3 cm are included in this study because PDAC risk with lesions less than 1 cm is quite low while lesions greater than 3 cm or with worrisome features by Fukuoka Consensus Guidelines have an appreciable risk of harboring an undiagnosed PDAC. All controls must have pancreatic imaging studies showing no evidence of PDAC within 6 months of sample collection.
  Interventions: Diagnostic Test: PancreaSure

INTERVENTIONS:
Diagnostic Test: PancreaSure — Serum-based biomarker test comprised of ELISA-based analyte readings of 4 protein biomarkers (ICAM-1, TIMP1, THSB1, and CTSD) and CA19-9 summed by a mathematical algorithm with associated coefficients where a pre-defined cutoff establishes a positive or negative detection of PDAC.

SUMMARY:
This is a case-control study to clinically validate the performance of PancreaSure, a protein biomarker test, to differentiate Stage I and Stage II pancreatic ductal adenocarcinoma (PDAC) patient samples from samples acquired from control patients not diagnosed with PDAC but at increased risk of disease due to familial/genetic history or clinical symptoms.

DETAILED DESCRIPTION:
This is the second case-control study to clinically validate the multi- analyte biomarker diagnostic model, PancreaSure. Serum samples will be collected for analysis from patients with pancreatic ductal adenocarcinoma (PDAC) Stages I and II and non-PDAC controls of similar demographics who were at increased risk of PDAC because of their familial or genetic history. Investigators and patients will not receive individual patient results, therefore patient care will not be impacted by test results. Analysis of blood samples will be conducted in Immunovia's laboratory in Durham, NC by personnel who are blinded to subject data. Biomarker results will be analyzed using a predefined (locked) algorithm with predefined (locked) cut-off resulting in a positive/negative test outcome.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent available
* > 45 years of age
* PDAC cases

  * Treatment-naïve, pathologically confirmed PDAC Stage I or Stage II
  * Sporadic or familial/genetic PDAC
* Controls

  * Individuals at high risk for PDAC because of their familial and/or genetic history
  * Individuals at high risk for PDAC because of pancreatic cysts between 1.0cm and 3.0cm in diameter.
  * Controls will be selected to have similar demographic features (age/gender) to PDAC patients

Exclusion Criteria:

* Prior treatment for PDAC (i.e., prior resection, radiotherapy, or chemotherapy)
* Current immunosuppressive (e.g., systemic steroid therapy) or chemotherapy
* Major surgery or significant trauma within 12 weeks prior to blood sample collection
* Non-PDAC malignancies within 3 years prior to sample collection squamous or basal cell skin carcinoma is not an exclusion criteria)
* Control patients who currently have

  * biliary obstruction secondary to gallstones
  * prior diagnosis or imaging evidence of chronic pancreatitis
  * cystic pancreatic lesions >3.0 cm in diameter or showing worrisome features according to Fukuoka Consensus Guidelines.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Samples will be retrospectively obtained under the Immunovia PanDetect, PanFam, or unique institutional protocols for sample collection through high-risk PDAC surveillance programs.
Sampling Method: Non-Probability Sample
Enrollment: 386 (Actual)
Dates: Start 2025-02-11 (Actual); Primary Completion 2025-03-24 (Actual); Study Completion 2025-04-07 (Actual)

PRIMARY OUTCOMES:
PancreaSure Sensitivity | Baseline
  Determine the sensitivity of PancreaSure in the classification of serum samples from patients diagnosed with PDAC as positive for PDAC, in a study sample containing both PDAC and control samples.

SECONDARY OUTCOMES:
PancreaSure Specificity | Baseline
  Determine specificity of PancreaSure in the classification of serum samples from control subjects as negative for PDAC, in a study sample containing both PDAC and control samples
Performance versus CA19-9 alone | Baseline
  Determine performance (sensitivity and specificity) of PancreaSure compared to CA19-9 alone in the overall population

CONTACTS AND LOCATIONS:
Overall Officials: Patricio Polanco, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (6):
- United States (6):
  - HonorHealth Clinical Research Institute, Scottsdale, Arizona
  - New York University Langone Health, New York, New York
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Regional One Health, Memphis, Tennessee
  - UT Southwestern Medical Center, Dallas, Texas
  - Virginia Commonwealth University, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No
Individual patient test results will not be shared with patients.